CLINICAL TRIAL: NCT01581437
Title: Recording for Potential AF Drivers and Patient Specific Atrial Anatomy and Atrial Electrogram Maps Using an FDA Approved 64-Pole Basket Catheter (CONFIRM)
Brief Title: Recording for Potential AF Drivers and Patient Specific Atrial Anatomy & Atrial Electrogram Maps
Acronym: CONFIRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: University of California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HM13720
Record Dates: First submitted 2012-04-06; First posted 2012-04-20 (Estimated); Results first posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; cardiac ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 64 pole basket catheter (Other): all patients participating undergo mapping using the 64 pole basket catheter to assess for Atypical areas of drivers that may cause atrial fibrillation
  Interventions: Procedure: 64 pole basket catheter

INTERVENTIONS:
Procedure: 64 pole basket catheter — The 64 pole basket catheter expands into a small flexible balloon that conforms to the atrial anatomy.
  Other Names: Constellation basket catheter

SUMMARY:
The 64 pole basket catheter used for the mapping procedure will be defined "atypical" sites which sustain atrial fibrillation. The ablation through the driver will lead to more rapid ablation of the atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a common abnormal and rapid heart rhythm characterized by erratic electrical activity of the upper chambers of the heart. This cardiac arrhythmia may lead to stroke, heart failure, low blood pressure, chest pain, and increased mortality rate. Treatment may include medication to stop the rhythm abnormality, blood thinners, and/or ablation. Ablation involves application of heat or freezing to the area sustaining the rhythm abnormality. This requires tubes (catheters)to be placed in the heart. Human atrial fibrillation may be sustained by localized drivers (rapid and/or organized sites of atrial electrical activation). By mapping/recording the patient's specific atrial anatomy and atrial electrical activity with the 64-pole basket catheter, we may add to the knowledge base of these driver locations. We may also add to the knowledge about where best to ablate to terminate the arrhythmia. Typical anatomic

ELIGIBILITY:
Inclusion Criteria:

* Patients at VCU Medical Center who are 21 years or older undergoing EPS for ablation of persistent AF (non-rheumatic) whose AF episodes last equal to or greater than 7 days but terminate with DC cardioversion or anti-arrhythmic drugs and do not recur within 24 hours.
* Per current standard of care, AF patients must have failed equal to or greater than 1 anti-arrhythmic drug to qualify for ablation.

Exclusion Criteria:

* Active coronary ischemic in the past year
* Rheumatic valve disease, that leads to distinct AF and increases thromboembolic risk
* Prior ablation or cardiac surgery, that alters atrial electophysiology
* Left atrial clot or dense contrast on TEE, which would increase thromboembolic risk
* Out of range serum electrolytes, including K outside 4.0-5.0 mmol/1
* Left atrial diameter greater than 60 mm, to exclude extreme structural remodeling and failure to maintain sinus rhythm
* Thrombotic disease, venous filters, transient ischemic attack or cerebrovascular accident, to minimize additional risk
* Pregnancy
* Inability or unwillingness to provide informed consent
* Unable to converse in English
* Use of anti-arrhythmic drug less than 5 X half-life Prior ablation or cardiac surgery, that alters atrial electophysiology

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Ellenbogen, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Result] Shivkumar K, Ellenbogen KA, Hummel JD, Miller JM, Steinberg JS. Acute termination of human atrial fibrillation by identification and catheter ablation of localized rotors and sources: first multicenter experience of focal impulse and rotor modulation (FIRM) ablation. J Cardiovasc Electrophysiol. 2012 Dec;23(12):1277-85. doi: 10.1111/jce.12000. Epub 2012 Nov 6. PMID 23130890
- [Result] Baykaner T, Clopton P, Lalani GG, Schricker AA, Krummen DE, Narayan SM; CONFIRM Investigators. Targeted ablation at stable atrial fibrillation sources improves success over conventional ablation in high-risk patients: a substudy of the CONFIRM Trial. Can J Cardiol. 2013 Oct;29(10):1218-26. doi: 10.1016/j.cjca.2013.07.672. Epub 2013 Aug 30. PMID 23993247

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 64 Pole Basket Catheter
Started | 78
Completed | 78
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 48 patients with persistent AF, 7=longstanding AF, 23 paroxysmal AF
Arm/Group | 64 Pole Basket Catheter
Number analyzed (Participants) | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 76
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 61 [48 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — specific numbers per gender not collected
  Male | NA — specific numbers per gender not collected
Region of Enrollment [Number; unit: participants]
  United States | 78
Atrial Fibrillation [Number; unit: participants] — Measure title Atrial Fibrillation
  participants
    persisitent atrial fibrillation | 48
    longstanding persisitent atrial fibrillation | 7
    paroxysmal atrial fibrillation | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Drivers in Right Atrial
Description: To determine where atypical areas of drivers might be.
Time Frame: 30 min
Measure: Number; unit: percentage of rotor sources
Arm/Group | 64 Pole Basket Catheter
Number analyzed (Participants) | 78
percentage of rotor sources | 25.3

2. Primary Outcome: Time to Ablation of All Sources
Description: total time taken to ablate all sources of rotors/focal sources in driver locations
Time Frame: 30 minutes
Population: patients participating undergo mapping using the 64 pole basket catheter
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- 64 Pole Basket Catheter: all patients participating undergo mapping using the 64 pole basket catheter to assess for Atypical areas of drivers that may cause atrial fibrillation
  64 pole basket catheter: The 64 pole basket catheter expands into a small flexible balloon that conforms to the atrial anatomy.
  Outcome:78 patients enrolled multicenter.
Arm/Group | 64 Pole Basket Catheter
Number analyzed (Participants) | 78
minutes | 16.6 (11.7)

3. Primary Outcome: Percentage of Patients With Greater Than One Right Atrial Source of Rotor/Focal Sources
Description: percentage of patients
Time Frame: 30 minutes
Measure: Number; unit: percentage of patients
Arm/Group | 64 Pole Basket Catheter
Number analyzed (Participants) | 78
percentage of patients | 50

4. Primary Outcome: Average Number of Rotors/Focal Drivers in Diverse Locations
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: rotor/focal drivers
Arm/Group | 64 Pole Basket Catheter
Number analyzed (Participants) | 78
rotor/focal drivers | 2.3 (0.9)

5. Secondary Outcome: Number of Participants With Successful Use of 64 Pole Basket Catheter at Non-University of California San Diego Electrophysiology Labs
Description: To determine if the 64 pole basket catheter will be successfully used to gather information on Atrial Fibrillation drivers.
Time Frame: 30 min
Measure: Number; unit: participants
Arm/Group | 64 Pole Basket Catheter
Number analyzed (Participants) | 78
participants | 78

6. Secondary Outcome: Mean Time to Recurrence of Atrial Fibrillation
Description: mean time to recurrence of atrial fibrillation
Time Frame: 1 year
Population: patients participating undergo mapping using the 64 pole basket catheter
Measure: Mean (Full Range); unit: days
Groups:
- 64 Pole Basket Catheter: all patients participating undergo mapping using the 64 pole basket catheter to assess for Atypical areas of drivers that may cause atrial fibrillation
  64 pole basket catheter: Outcome:78 patients enrolled multicenter
Arm/Group | 64 Pole Basket Catheter
Number analyzed (Participants) | 78
days | 245 [0 to 365]

7. Secondary Outcome: Single-procedure Freedom From Atrial Fibrillation
Description: percentage of patients without prior ablation
Time Frame: one year
Population: percentage of patients who underwent mapping with 64 pole basket catheter
Measure: Number; unit: percentage of patients with no prior abl
Groups:
- 64 Pole Basket Catheter: all patients participating undergo mapping using the 64 pole basket catheter to assess for Atypical areas of drivers that may cause atrial fibrillation
  64 pole basket catheter:
Arm/Group | 64 Pole Basket Catheter
Number analyzed (Participants) | 78
percentage of patients with no prior abl | 87.5

8. Secondary Outcome: Percentage of All Patients Who Underwent Ablation of Rotor/Focal Sources of Atrial Fibrillation
Description: percentage of all patients who had ablation perfornmed
Time Frame: 1 year
Population: all patients participating undergo mapping using the 64 pole basket catheter
Measure: Number; unit: percentage of all patients undergoing ab
Arm/Group | 64 Pole Basket Catheter
Number analyzed (Participants) | 78
percentage of all patients undergoing ab | 80.5

ADVERSE EVENTS:
Arm/Group | 64 Pole Basket Catheter
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No